CLINICAL TRIAL: NCT04164719
Title: A Single-dose, Randomized, Open-label, 3-way Crossover Study to Evaluate the Dose-proportionality and Food Effect of TNX-102 SL (Cyclobenzaprine HCl Sublingual Tablets) in Healthy Subjects
Brief Title: Dose-Proportionality and Food Effect Study of TNX-102 SL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tonix Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TNX-CY-F110
Record Dates: First submitted 2019-11-13; First posted 2019-11-15 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — cyclobenzaprine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A (Experimental): TNX-102 SL 2.8 mg, under fasting conditions
  Interventions: Drug: TNX-102 SL
- Treatment B (Experimental): TNX-102 SL 5.6 mg (2 x 2.8 mg sublingual tablets), under fasting conditions
  Interventions: Drug: TNX-102 SL
- Treatment C (Experimental): TNX-102 SL 5.6 mg (2 x 2.8 mg sublingual tablets), under fed conditions
  Interventions: Drug: TNX-102 SL

INTERVENTIONS:
Drug: TNX-102 SL — Subjects will place TNX-102 SL sublingual tablets under the tongue until dissolved, and not to crush or chew them
  Other Names: cyclobenzaprine HCl

SUMMARY:
This will be a single center, single-dose, randomized, open-label, 3-period, crossover, dose-proportionality and food-effect study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, non-smoker, ≥18 and ≤65 years of age, with Body Mass Index (BMI) >18.5 and <30.0 kg/m2
* Females of childbearing potential must be willing to use a medically acceptable method of birth control throughout the study
* Capable of consent

Exclusion Criteria:

* Any clinically significant abnormality or abnormal laboratory test results found during medical screening
* Positive hepatitis B, hepatitis C, HIV, urine drug screen, urine cotinine test, or alcohol breath test at screening
* History of allergic reactions to cyclobenzaprine, any of the formulation components, or other related drugs
* Use of any drugs known to induce or inhibit hepatic drug metabolism within 30 days prior to the first study drug administration
* Positive pregnancy test at screening
* Clinically significant electrocardiogram (ECG) abnormalities or vital sign abnormalities at screening
* History of significant alcohol or drug abuse within one year prior to screening
* Participation in a clinical trial involving the administration of an investigational or marketed drug within 30 days prior to the first dosing or concomitant participation in an investigational study involving no drug administration
* Use of medication other than topical products without significant systemic absorption and hormonal contraceptives
* Donation of plasma within 7 days prior to dosing, or significant loss of blood within 54 days of dosing.
* Abnormal hemoglobin and hematocrit levels at screening
* Breast-feeding subject
* Presence of orthodontic braces or orthodontic retention wires, or any physical findings in the mouth or tongue that would be likely to interfere with successful completion of the dosing procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2019-12-24 (Actual); Study Completion 2019-12-24 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration Versus Time Curve (AUC) of TNX-102 SL 5.6 mg versus TNX-102 SL 2.8 mg under fasting conditions | Day 1 to Day 6
  Blood samples are collected from pre-dose on Day 1 up until Day 6 (144 hours post-dose)
Area Under the Plasma Concentration Versus Time Curve (AUC) of TNX-102 SL 5.6 mg versus TNX-102 SL 5.6 mg under fed conditions | Day 1 to Day 6
  Blood samples are collected from pre-dose on Day 1 up until Day 6 (144 hours post-dose)
Number of Subjects With Treatment-Emergent Adverse Events (TEAEs) of TNX-102 SL 2.8 mg versus TNX-102 SL 5.6 mg under fasting conditions | Day 1 to Day 15
  Blood samples are collected from pre-dose on Day 1 up until Day 15 (360 hours post-dose)
Number of Subjects With Treatment-Emergent Adverse Events (TEAEs) of TNX-102 SL 5.6 mg under fasted and fed conditions | Day 1 to Day 15
  Blood samples are collected from pre-dose on Day 1 up until Day 15 (360 hours post-dose)

CONTACTS AND LOCATIONS:
Overall Officials: Denis Audet, MD, Principal Investigator — Contract Research Organization
Locations (1):
- Canada, Quebec, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No